CLINICAL TRIAL: NCT05430373
Title: A Single-arm Phase I Clinical Study of GT101 Injection for the Treatment of Metastatic or Recurrent Solid Tumors
Brief Title: GT101 Injection for the Treatment of Metastatic or Recurrent Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Grit Biotechnology (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GT101-101
Record Dates: First submitted 2022-06-13; First posted 2022-06-24 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Solid Tumors, Adult

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- GT101 treatment group (Other): Autologous tumor infiltrating lymphocyte injection
  Interventions: Biological: GT101

INTERVENTIONS:
Biological: GT101 — Autologous tumor infiltrating lymphocyte injection

SUMMARY:
This is a multicenter, single-arm phase I clinical trial.The study process was divided into: screening period, sampling and production period, lymphodepleting chemotherapy period, treatment and observation period, and follow-up period.

The study is designed to enroll 20-31 subjects, with 14-20 subjects expected to be evaluable, in an "autologous tumor-infiltrating lymphocyte therapy" regimen that includes：

1. Clear lymphatic pretreatment (FC regimen: cyclophosphamide + fludarabine).
2. GT101 infusion.
3. post-infusion treatment (interleukin-2 intravenous push).

ELIGIBILITY:
Inclusion Criteria:

* 1. The Patients (or legally authorized representative) Patients (or legally authorized representative) must have the ability to understand the requirements of the study, have provided written informed consent as evidenced by signature on an informed consent form (ICF) approved by an Institutional Review Board/Independent Ethics Committee (IRB/IEC), must have the ability to understand the requirements of the study;
* 2.Must have a confirmed diagnosis of malignancy of their receptive histologies or cytologies: unresectable recurrent or metastatic solid tumor;
* 3.At least one resectable lesion (preferably superficial metastatic lymph nodes) that has not been treated with radiation and has not received other local therapies. The separated tissues mass weighing ≥1.0g (either of single lesion origin or multiple lesions combined) for the preparation of autologous tumor-infiltrating lymphocytes. Minimally invasive treatment where possible;

Exclusion Criteria:

* 1. Patients who have symptomatic and/or untreated CNS metastases (Except stable brain metastases, no medication required within 3 months, no hormone dependence);
* 2.The patient who has any active autoimmune disease, history of autoimmune disease, need for systemic steroid hormones or a condition requiring immunosuppressive drug therapy (>10 mg/day of prednisone or equivalent hormone);
* 3. Arterial/venous thrombotic events within 6 months prior to surgical operation, such as: cerebrovascular accident, deep vein thrombosis and pulmonary embolism occurring;
* 4.Active infections requiring treatment with systemic anti-infectives (except for topical antibiotics); or those with unexplained fever > 38.5℃ occurring during the screening period, except for tumor fever;
* 5. Patients who have refractory or intractable epilepsy, poorly controlled hydrothorax, hydrops abdominis, active gastrointestinal bleeding or IL-2 contraindications;
* 6. Participate in other clinical trials within 28 days prior to the first dose of this study, or planning to participate in this study and other clinical trials at the same time;
* 7. Patients who have received allogeneic bone marrow transplantation or an organ allograft;
* 8.Patients who have a history of hypersensitivity to any component or excipient of study drugs: autologous tumor infiltrating lymphocytes, cyclophosphamide, fludarabine, IL-2, dimethyl sulfoxide (DMSO), human serum albumin (HSA), dextran-40 and antibiotics (beta lactam antibiotics, gentamicin);

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2022-05-23 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety Profile Measured by Grade ≥3 TEAEs | 3 years
  To characterize the safety profile of autologous TIL injection（GT101) in patients with relapsed/metastatic advanced solid tumor as measured by the incidence of Grade ≥ 3 treatment-emergent adverse events (TEAEs)
Objective response rate | 3 years
  To evaluate efficacy parameters such Objective Response Rate (ORR) per RECIST 1.1, as assessed by the Investigator
Overall survival | 3 years
  To evaluate efficacy parameters such Overall Survival (OS)
Progression-free survival | 3 years
  To evaluate efficacy parameters such Progression-Free Survival (PFS) per RECIST 1.1, as assessed by the Investigator
Disease Control Rate | 3 years
  To evaluate efficacy parameters such disease control rate (DCR) per RECIST 1.1, as assessed by investigater
Duration of Response | 3 years
  To evaluate efficacy parameters such duration of response (DoR) per RECIST 1.1, as assessed by investigater

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - The fifth medical center of the General Hospital of the Chinese people's Liberation Army, Beijing, Beijing Municipality
  - Chongqing University Cancer Center, Chongqing, Chongqing Municipality
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - West China School of Medicine/West China Hospital of Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No